CLINICAL TRIAL: NCT07389031
Title: Maralixibat for the trEatment of inTrAhePatic cHOlestasis of pRegnancy (METAPHOR)
Brief Title: Maralixibat for Intrahepatic Cholestasis of Pregnancy
Acronym: METAPHOR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1012589; X (Other Grant/Funding Number: Mirum Pharmaceuticals, Inc.)
Record Dates: First submitted 2026-01-26; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: Pruritus; Itch; Itching; Cholestasis; Bile Acid; Pregnancy; Pregnant; Intrahepatic; Liver
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Pruritus; Cholestasis | interventions — maralixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Maralixibat (Experimental): Dose-titrated open-label maralixibat, with primary assessment at Week 3; participants may continue treatment until delivery
  Interventions: Drug: Maralixibat

INTERVENTIONS:
Drug: Maralixibat — Oral solution, dose-titrated. Maralixibat is an ileal bile acid transporter (IBAT) inhibitor.

SUMMARY:
An open label phase 2a/b trial of maralixibat in patients with Intrahepatic Cholestasis of Pregnancy (ICP) and elevated serum bile acid concentrations (sBA) to evaluate safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent and be willing to comply with all study visits and requirements through end of study, including the follow-up period
2. Female aged ≥18 and ≤50 years with a viable singleton pregnancy between 20 weeks 0 days and 34 weeks 0 days (inclusive) at the screening visit, and no more than 35 weeks 0 days (inclusive) at the baseline visit.
3. Diagnosis of ICP
4. Non fasting (e.g., postprandial) tSBA level ≥19 μmol/L as assessed by the local laboratory.
5. Meets all inclusion criteria and no exclusion criteria at screening as well as at the Day 1 (baseline) visit, unless otherwise specified.

Exclusion Criteria:

1. At the time of either the screening or baseline visit, decision has already been made to deliver within the next 7 days, for any indication.
2. Known non-reassuring fetal status based upon antepartum testing (e.g., NST/CTG) at or within 7 days before the baseline visit.
3. Known fetal anomaly likely to result in intrauterine fetal demise or neonatal death within the first 30 days of life.
4. Participating in another ongoing interventional clinical study at screening or planning to participate in another contemporaneous interventional clinical study while participating in this study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Assess the Safety and Tolerability of Maralixibat in Participants With ICP | Through to end of treatment, up to 21 weeks
  To assess the safety and tolerability of maralixibat in participants with ICP on the basis of the following endpoints:
  Proportion of participants experiencing one or more of the following:
  To assess the safety and tolerability of maralixibat for the treatment of intrahepatic cholestasis of pregnancy (ICP) in pregnant women.
  Incidence of adverse events (AEs), serious adverse events (SAEs), and AEs that lead to discontinuation
  Incidence of clinically relevant laboratory abnormalities .

SECONDARY OUTCOMES:
Mean Change in the Weekly Average Worst Daily Itch Score as Measured by the Adult Itch Reported Outcome (5-D Itch Scale) | Through the end of treatment (up to 21 weeks).
  Mean change from baseline to Week 3 (minimum 7 days) of the study treatment period in the weekly average worst daily itch score as measured by the Adult Itch Reported Outcome (5-D Itch Scale)
Mean Change in Total Serum Bile Acid (tSBA) Concentration | Baseline to Week 3 (minimum 7 days of treatment)
  Mean change from baseline to Week 3 of the study treatment period in total tSBA concentration (minimum 7 days).

OTHER OUTCOMES:
Proportion of participants with a Composite Adverse Perinatal Outcome | Up to 28 days after delivery
  Number of adverse outcomes recorded from baseline to birth visit/end of study

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Williamson, MD, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Birmingham Womens and Childrens NHS Foundation Trust, Birmingham
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No